CLINICAL TRIAL: NCT00525174
Title: A Randomized Trial of Full-time Bangerter Filters Versus Part-time Daily Patching for the Treatment of Moderate Amblyopia in Children
Brief Title: Full-time Bangerter Filters Versus Part-time Daily Patching for Moderate Amblyopia in Children
Acronym: ATS10
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Ray Kraker, Director, PEDIG Coordinating Center, Jaeb Center for Health Research
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEI-136; 2U10EY011751 (NIH)
Record Dates: First submitted 2007-08-31; First posted 2007-09-05 (Estimated); Results first posted 2011-06-17 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Amblyopia
Keywords: Amblyopia; Patching; Bangerter filters
MeSH Terms: conditions — Amblyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patching (Active Comparator): 2 hours daily patching of the sound eye plus one hour near activities while patching
  Interventions: Device: Patching; Procedure: Near activities
- Bangerter filters (Active Comparator): Bangerter filter worn on sound eye spectacles lens full time plus at least one hour near activities
  Interventions: Device: Bangerter filters; Procedure: Near activities

INTERVENTIONS:
Device: Bangerter filters — Bangerter filter worn on sound eye spectacle lens full time
  Arms: Bangerter filters
Device: Patching — 2 hours daily patching of the sound eye
  Other Names: Coverlet, 3M Opticlude, Ortopad®
  Arms: Patching
Procedure: Near activities — one hour near visual activities

SUMMARY:
This study is a randomized clinical trial designed to evaluate the non-inferiority of Bangerter filters compared to 2 hours of daily patching as a primary treatment for moderate amblyopia (20/40 to 20/80) in children ages 3 to < 10 years.

Secondary objectives of this study are (1) to determine the time course of visual improvement with Bangerter filter treatment, (2) to compare patient quality of life, measured by a modified Amblyopia Treatment Index, between patients treated with patching vs. Bangerter filters, (3) to determine whether blurring the sound eye to a visual acuity worse than the amblyopic eye predicts improvement in acuity, and (4) to determine whether a change in fixation to the amblyopic eye is predictive of improvement in visual acuity.

The primary outcome assessment is visual acuity at 24 weeks for both the amblyopic and sound eyes.

The primary analytic approach for the amblyopic eye acuity will involve construction of a one-sided 95% confidence interval to assess non-inferiority based on a treatment group comparison of logMAR visual acuity scores adjusted for baseline visual acuity scores in an analysis of covariance (ANCOVA) model.

Sound eye acuity data will be reported for each treatment regimen at the 24-week visit as mean change (logMAR lines) from baseline and as the distribution of the number of lines of change from baseline.

DETAILED DESCRIPTION:
Amblyopia is the most common cause of monocular visual impairment in children, estimated to affect as many as 3.6% of the childhood population. The natural history of amblyopia is relatively unknown although it has been reported that visual acuity may deteriorate further without treatment.

Although occlusion or patching of the sound eye has been the mainstay for amblyopia therapy, alternative treatment such as pharmacological or optical penalization may be as effective. In a randomized, controlled clinical trial of 419 children, 3 years to less than 7 years old with moderate amblyopia, patching was compared to atropine. Although improvement with atropine was initially slower, both treatments produced similar improvement after 6 months.

Although both patching and atropine have been proven effective for treating amblyopia, neither treatment is without adverse side effects. Patching is associated with compliance difficulties, the need for continuous monitoring, and social stigma. Negative side effects observed in children treated with atropine include light sensitivity, facial flushing, and fever. In a randomized clinical trial comparing patching to atropine as a treatment for amblyopia, a questionnaire to assess the impact of patching and atropine treatment on the child and family indicated that both treatments were well tolerated overall, however, patching had lower compliance and higher social stigma than atropine.

Bangerter filters, also known as Bangerter foils, have been used mainly as secondary amblyopia therapy following patching or atropine to either further improve or maintain the visual gain. One advantage of Bangerter filters compared to patching is that the lower density filters are not readily apparent and therefore would be expected to increase patient compliance due to reduced social stigma. Another advantage of Bangerter filters is that there is no opportunity for skin irritation from bandage adhesive, a commonly-reported side effect of patching. In addition, there is a theoretical advantage that Bangerter filters are less disruptive to binocular function during treatment compared to other modalities such as patching.

Few data are available comparing Bangerter filters with patching for the treatment of amblyopia. Bonsall randomized 14 patients, 3 to 10 years old, with previously untreated strabismic/anisometropic amblyopia to either 6 hours of daily patching or full-time Bangerter filters. Baseline amblyopic eye acuity was 20/30 to 20/400 for the patching group and 20/30 to 20/200 for the Bangerter group. The Bangerter filter prescribed was the minimum density foil needed to elicit a switch in fixation from the sound eye to the amblyopic eye. Visual acuity was measured every 6-8 weeks until the amblyopic eye visual acuity was equal to that of the sound eye, an improvement that was achieved in 5 of the 14 at the time the study was stopped. The average time to achieve equal vision between the amblyopic and sound eyes was about 4.5 months (142 days) for the foil group versus about 9 months (272 days) for the patching group. Both forms of therapy were equally tolerated. Despite good preliminary data, a large randomized clinical trial comparing the effectiveness of Bangerter filters to patching for the treatment of amblyopia has yet to be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Age 3 to < 10 years
* Amblyopia associated with strabismus, anisometropia, or both
* No ocular cause apparent for reduced visual acuity
* Visual acuity 20/40 to 20/80 (71 to 54 letters inclusive) in amblyopic eye
* Visual acuity 20/40 or better (>= 69 letters) in sound eye
* Interocular difference >= 3 logMAR lines (>= 15 letters)
* No amblyopia treatment other than spectacles in last 6 months

  *Any treatment more than 6 months prior to enrollment is acceptable
* Currently wearing spectacles
* Appropriate spectacles have been worn for 16 weeks prior to enrollment or visual acuity documented to be stable
* No myopia > -6.00 D spherical equivalent in either eye
* Cycloplegic refraction within 6 months prior to enrollment
* Ocular examination within 6 months prior to enrollment

Exclusion Criteria:

* Current vision therapy or orthoptics
* Ocular cause for reduced visual acuity
* Prior intraocular or refractive surgery
* Known skin reactions to patch or bandage adhesives

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 186 (Actual)
Dates: Start 2007-11; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert P. Rutstein, O.D., M.S., Study Chair — University of Alabama at Birmingham; Graham E. Quinn, M.D., MSCE, Study Chair — Children's Hospital of Philadelphia
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Result] Pediatric Eye Disease Investigator Group Writing Committee; Rutstein RP, Quinn GE, Lazar EL, Beck RW, Bonsall DJ, Cotter SA, Crouch ER, Holmes JM, Hoover DL, Leske DA, Lorenzana IJ, Repka MX, Suh DW. A randomized trial comparing Bangerter filters and patching for the treatment of moderate amblyopia in children. Ophthalmology. 2010 May;117(5):998-1004.e6. doi: 10.1016/j.ophtha.2009.10.014. Epub 2010 Feb 16. PMID 20163869
- [Result] Rutstein RP, Foster NC, Cotter SA, Kraker RT, Lee DH, Melia M, Quinn GE, Tamkins SM, Wallace DK; Pediatric Eye Disease Investigator Group. Visual acuity through Bangerter filters in nonamblyopic eyes. J AAPOS. 2011 Apr;15(2):131-4. doi: 10.1016/j.jaapos.2010.11.015. Epub 2011 Mar 21. PMID 21419678
- [Derived] Wallace DK, Lazar EL, Melia M, Birch EE, Holmes JM, Hopkins KB, Kraker RT, Kulp MT, Pang Y, Repka MX, Tamkins SM, Weise KK; Pediatric Eye Disease Investigator Group. Stereoacuity in children with anisometropic amblyopia. J AAPOS. 2011 Oct;15(5):455-61. doi: 10.1016/j.jaapos.2011.06.007. PMID 22108357

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligibility criteria included age 3 to <10 years, visual acuity in the amblyopic eye 20/40 to 20/80, fellow eye visual acuity of 20/40 or better, interocular acuity difference of 3 or more lines, and the presence or history of strabismus and/or anisometropia.
Pre-assignment Details: At enrollment, subjects were required to have been wearing spectacles with optimal correction for a minimum of 16 weeks or until stability of visual acuity was documented (no improvement in amblyopic visual acuity at 2 consecutive visits at least 4 weeks apart).
Period: Overall Study
Arm/Group | Patching | Bangerter Filters
Started | 97 | 89
Completed | 88 | 81
Not Completed | 9 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patching | Bangerter Filters | Total
Number analyzed (Participants) | 97 | 89 | 186
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.3 (1.62) | 6.3 (1.67) | 6.3 (1.64)
Age, Customized [Number; unit: participants] — Age at enrollment in years
  participants
    3 to <7 years | 62 | 57 | 119
    7 to <10 years | 35 | 32 | 67
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 36 | 84
  Male | 49 | 53 | 102
Race/Ethnicity, Customized [Number; unit: participants]
  White | 67 | 69 | 136
  African-American | 13 | 1 | 14
  Hispanic or Latino | 11 | 15 | 26
  Asian | 3 | 0 | 3
  More than 1 race | 2 | 3 | 5
  Unknown / not reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 97 | 89 | 186
Prior treatment for amblyopia at enrollment [Number; unit: participants]
  None | 83 | 72 | 155
  Patching | 8 | 5 | 13
  Atropine | 2 | 3 | 5
  Patching and atropine | 4 | 9 | 13
Cause of amblyopia [Number; unit: participants]
  Strabismus | 27 | 23 | 50
  Anisometropia | 42 | 39 | 81
  Strabismus and anisometropia | 28 | 27 | 55
Distance visual acuity in amblyopic eye [Number; unit: participants] — Visual acuity was measured in each eye using the Amblyopia Treatment Study (ATS) visual acuity testing protocol resulting in a Snellen acuity score that can range from 20/16 to 20/800 for ages 3 to <7; or with the electronic early treatment diabetic retinopathy study (E-ETDRS) method for 7 to <10 year olds which resulted in a letter score that could range from 0 to 97 letters, with 0 being the worst and 97 being the best. Scores were converted to log of minimum angle of resolution (logMAR) equivalents for analyses (lower logMAR value is better than higher logMAR).
  participants
    20/80 (0.62 - 0.56 logMAR) (worse) | 23 | 16 | 39
    20/63 (0.54 - 0.46 logMAR) | 31 | 27 | 58
    20/50 (0.44 - 0.36 logMAR) | 22 | 24 | 46
    20/40 (0.34 - 0.28 logMAR) (best) | 21 | 22 | 43
Mean (SD) Distance Visual Acuity in Amblyopic Eye [Mean (Standard Deviation); unit: logMAR] — Visual acuity was measured in each eye using the Amblyopia Treatment Study (ATS) visual acuity testing protocol resulting in a Snellen acuity score that can range from 20/16 to 20/800 for ages 3 to <7; or with the electronic early treatment diabetic retinopathy study (E-ETDRS) method for 7 to <10 year olds which resulted in a letter score that could range from 0 to 97 letters, with 0 being the worst and 97 being the best. Scores were converted to log of minimum angle of resolution (logMAR) equivalents for analyses (lower logMAR value is better than higher logMAR).
  logMAR | 0.46 (0.10) | 0.44 (0.10) | 0.45 (0.10)
Distance visual acuity in fellow eye [Number; unit: participants] — Visual acuity was measured with the Amblyopia Treatment Study single-surround HOTV (ATS-HOTV) method for subjects aged 3 to <7 years or the Electronic Early Treatment Diabetic Retinopathy Study (E-ETDRS) method for subjects aged 7 to <10 years.
  participants
    20/40 (0.32 to 0.26 logMAR) (worse) | 2 | 3 | 5
    20/32 (0.24 to 0.16 logMAR) | 16 | 9 | 25
    20/25 (0.14 to 0.06 logMAR) | 17 | 19 | 36
    20/20 (0.04 to -0.04 logMAR) | 42 | 40 | 82
    20/16 (-0.06 to -0.14 logMAR) (best) | 20 | 18 | 38
Mean (SD) Distance Visual Acuity in Fellow Eye [Mean (Standard Deviation); unit: logMAR] — Visual acuity was measured in each eye using the Amblyopia Treatment Study (ATS) visual acuity testing protocol resulting in a Snellen acuity score that can range from 20/16 to 20/800 for ages 3 to <7; or with the electronic early treatment diabetic retinopathy study (E-ETDRS) method for 7 to <10 year olds which resulted in a letter score that could range from 0 to 97 letters, with 0 being the worst and 97 being the best. Scores were converted to log of minimum angle of resolution (logMAR) equivalents for analyses (lower logMAR value is better than higher logMAR).
  logMAR | 0.04 (0.10) | 0.03 (0.10) | 0.04 (0.10)
Intereye acuity difference [Mean (Standard Deviation); unit: logMAR line] — The difference between eyes in logMAR acuity was calculated with positive values indicating sound eye better. One letter = .02 logMAR, .1 logMAR = 5 letters or one line of visual acuity.
  logMAR line | 4.2 (1.1) | 4.1 (1.1) | 4.1 (1.1)
Spherical equivalent in amblyopic eye [Number; unit: diopter] — Spherical equivalent in diopters defined from cycloplegic refraction as sphere plus half the cylinder value
  diopter
    <0.00 | 3 | 8 | 11
    0 to < +1.00 | 2 | 2 | 4
    +1.00 to < +2.00 | 8 | 1 | 9
    +2.00 to < +3.00 | 6 | 10 | 16
    +3.00 to < +4.00 | 10 | 13 | 23
    >= +4.00 | 68 | 55 | 123
Mean (SD) spherical equivalent in amblyopic eye [Mean (Standard Deviation); unit: diopter] — Spherical equivalent in diopters defined from cycloplegic refraction as sphere plus half the cylinder value.
  diopter | 4.41 (2.21) | 4.15 (2.57) | 4.29 (2.38)
Spherical equivalent in fellow eye [Number; unit: diopter] — Spherical equivalent in diopters defined from cycloplegic refraction as sphere plus half the cylinder value
  diopter
    <0.00 | 1 | 5 | 6
    0 to < +1.00 | 18 | 16 | 34
    +1.00 to < +2.00 | 25 | 21 | 46
    +2.00 to < +3.00 | 13 | 12 | 25
    +3.00 to < +4.00 | 8 | 13 | 21
    >= +4.00 | 32 | 22 | 54
Mean (SD) spherical equivalent in fellow eye [Mean (Standard Deviation); unit: diopter] — Spherical equivalent in diopters defined from cycloplegic refraction as sphere plus half the cylinder value.
  diopter | 2.81 (2.14) | 2.49 (2.13) | 2.66 (2.14)

OUTCOME MEASURES:

1. Primary Outcome: Distribution of Visual Acuity in the Amblyopic Eye at 24 Weeks
Description: Visual acuity was measured in each eye using the Amblyopia Treatment Study (ATS) visual acuity testing protocol resulting in a Snellen acuity score that can range from 20/16 to 20/800 for ages 3 to <7; or with the electronic early treatment diabetic retinopathy study (E-ETDRS) method for 7 to <10 year olds which resulted in a letter score that could range from 0 to 97 letters, with 0 being the worst and 97 being the best. Scores were converted to log of minimum angle of resolution (logMAR) equivalents for analyses (lower logMAR value is better than higher logMAR).
Time Frame: 24 weeks
Measure: Number; unit: participants
Arm/Group | Bangerter | Patching
Number analyzed (Participants) | 81 | 88
participants
  20/125 (0.84 to 0.76 logMAR) (worse) | 1 | 0
  20/100 (0.74 to 0.66 logMAR) | 3 | 0
  20/80 (0.64 to 0.56 logMAR) | 3 | 1
  20/63 (0.54 to 0.46 logMAR) | 7 | 8
  20/50 (0.44 to 0.36 logMAR) | 5 | 12
  20/40 (0.34 to 0.26 logMAR) | 19 | 19
  20/32 (0.24 to 0.16 logMAR) | 14 | 20
  20/25 (0.14 to 0.06 logMAR) | 20 | 17
  20/20 (0.04 to -0.04 logMAR) | 9 | 7
  20/16 (-0.06 to -0.14 logMAR) (best) | 0 | 4

2. Primary Outcome: Mean (SD) of Amblyopic Eye Visual Acuity at 24 Weeks
Description: as for outcome 1
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Bangerter | Patching
Number analyzed (Participants) | 81 | 88
logMAR | 0.25 (0.19) | 0.23 (0.16)

3. Primary Outcome: Distribution of Change in Amblyopic Eye Visual Acuity Scores From Baseline to 24 Weeks
Description: Visual acuity was measured in each eye using the Amblyopia Treatment Study (ATS) testing protocol resulting in a Snellen acuity score for 3 to <7 year olds; or with the electronic early treatment diabetic retinopathy study (E-ETDRS) method for 7 to <10 year olds, resulting in a letter score that could range from 0 to 97 letters (0 worst; 97 best). Scores were converted to log of minimum angle of resolution (logMAR)(lower logMAR indicates better score). 'Worse' indicates acuity at 24 weeks is worse than acuity at baseline; 'Better' indicates acuity at 24 weeks is better than acuity at baseline.
Time Frame: Baseline to 24 weeks
Measure: Number; unit: participants
Arm/Group | Bangerter | Patching
Number analyzed (Participants) | 81 | 88
participants
  >= 3 lines worse | 1 | 0
  2 lines worse | 2 | 0
  1 line worse | 5 | 1
  0 lines | 8 | 4
  1 line better | 12 | 19
  2 lines better | 20 | 27
  >=3 lines better | 33 | 37
Statistical Analysis 1: Comparison: Bangerter vs Patching; Logistic regression was performed comparing the proportions of patients in each treatment group who had no improvement or worsening in amblyopic eye visual acuity from baseline to 24 weeks (change from baseline <= +4 letters for E-ETDRS testing); Test type: Superiority or Other; p = 0.02, Regression, Logistic

4. Primary Outcome: Mean Change in Amblyopic Eye Visual Acuity From Baseline to 24 Weeks
Description: Visual acuity was measured in each eye using the Amblyopia Treatment Study (ATS) testing protocol resulting in a Snellen acuity score for 3 to <7 year olds; or with the electronic early treatment diabetic retinopathy study (E-ETDRS) method for 7 to <10 year olds, resulting in a letter score that could range from 0 to 97 letters (0 worst; 97 best). Scores were converted to log of minimum angle of resolution (logMAR)(lower logMAR indicates better score). Change from baseline to 24 weeks was calculated. A positive difference indicates improvement (one logMAR line = 5 letters or one Snellen line).
Time Frame: Baseline to 24 weeks
Measure: Mean (Standard Deviation); unit: logMAR line
Arm/Group | Bangerter | Patching
Number analyzed (Participants) | 81 | 88
logMAR line | 1.9 (1.6) | 2.3 (1.3)
Statistical Analysis 1: Comparison: Bangerter vs Patching; The trial was designed as a non-inferiority study. The sample size was computed to be 170 subjects to have 90% power and a type I error rate of 5% for a noninferiority limit of 0.075 logarithm of minimum angle of resolution (logMAR), based on assumed standard deviation of 24-week visual acuity scores of 0.16 logMAR, a correlation between baseline and final acuities of 0.20, and 10% noncompletion of the study primary outcome examination; Test type: Non-Inferiority or Equivalence — The trial was designed as a non-inferiority study. The sample size was computed to be 170 subjects to have 90% power and a type I error rate of 5% for a noninferiority limit of 0.075 logarithm of minimum angle of resolution (logMAR), based on assumed standard deviation of 24-week visual acuity scores of 0.16 logMAR, a correlation between baseline and final acuities of 0.20, and 10% noncompletion of the study primary outcome examination; ANCOVA; The logMAR visual acuity scores were adjusted for baseline amblyopic eye acuity; Mean Difference (Net) = 0.38, 95% CI 1-sided [upper limit 0.76]
Statistical Analysis 2: Comparison: Bangerter vs Patching; In addition to the test of non-inferiority, an efficacy test of Patching over Bangerter filters was also completed; Test type: Superiority or Other; p = 0.09, ANCOVA; The logMAR visual acuity scores were adjusted for baseline amblyopic eye acuity; Mean Difference (Net) = 0.38, 95% CI 2-sided [-0.06 to 0.83]
Statistical Analysis 3: Comparison: Bangerter vs Patching; Treatment group difference in rate of improvement was evaluated using a population averaged linear mixed model after performing an inverse transformation of time to obtain linearity; Test type: Superiority or Other; p = 0.20, Mixed Models Analysis
Statistical Analysis 4: Comparison: Bangerter; The relationship between the fellow eye blur from the Bangerter filter at baseline and amblyopic improvement at the 24-week outcome was evaluated with an ANCOVA model with acuity in the fellow eye being categorized as better than versus equal to or worse than acuity in the amblyopic eye; Test type: Superiority or Other; p = 0.49, ANCOVA
Statistical Analysis 5: Comparison: Bangerter; The association of fixation preference while the Bangerter filter was over the fellow eye at baseline (amblyopic eye, fellow eye, alternates) with 24-week amblyopic eye acuity was evaluated in an ANCOVA model; Test type: Superiority or Other; p = 0.21, ANCOVA

5. Secondary Outcome: Mean Interocular Difference at 24 Weeks
Description: Visual acuity was measured in each eye using the Amblyopia Treatment Study (ATS) testing protocol resulting in a Snellen acuity score for 3 to <7 year olds; or with the electronic early treatment diabetic retinopathy study (E-ETDRS) method for 7 to <10 year olds, resulting in a letter score that could range from 0 to 97 letters (0 worst; 97 best). Scores were converted to log of minimum angle of resolution (logMAR)(lower logMAR indicates better score). A positive interocular difference indicates worse acuity in the amblyopic eye (one logMAR line = 5 letters or one Snellen line).
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: logMAR line
Arm/Group | Bangerter | Patching
Number analyzed (Participants) | 81 | 88
logMAR line | 2.3 (2.0) | 2.3 (1.5)

6. Secondary Outcome: Distribution of Subjects With Interocular Difference <1 logMAR Line at 24 Weeks
Description: as for outcome 5
Time Frame: 24 weeks
Measure: Number; unit: participants
Arm/Group | Bangerter | Patching
Number analyzed (Participants) | 81 | 87
participants | 15 | 10
Statistical Analysis 1: Comparison: Bangerter vs Patching; Logistic regression was used to compare the proportion of patients in each treatment group with amblyopic eye visual acuity within 1 line of the fellow eye or better; Test type: Superiority or Other; p = 0.27, Regression, Logistic

7. Secondary Outcome: Distribution of Subjects With >= 20/25 Amblyopic Eye Visual Acuity at 24 Weeks
Description: as for outcome 1
Time Frame: 24 weeks
Measure: Number; unit: participants
Arm/Group | Bangerter | Patching
Number analyzed (Participants) | 81 | 87
participants | 29 | 27
Statistical Analysis 1: Comparison: Bangerter vs Patching; Logistic regression was used to compare the proportion of patients in each treatment group with amblyopic visual acuity 20/25 or better at 24 weeks; Test type: Superiority or Other; p = 0.86, Regression, Logistic
Statistical Analysis 2: Comparison: Bangerter vs Patching; The time to first achieve amblyopic eye visual acuity of 20/25 or better was evaluated using a Cox proportional hazard model; Test type: Superiority or Other; p = 0.28, Regression, Cox

8. Secondary Outcome: Distribution of Subjects With 3 or More Lines of Improvement
Description: as for outcome 4
Time Frame: Baseline to 24 weeks
Measure: Number; unit: participants
Arm/Group | Bangerter | Patching
Number analyzed (Participants) | 81 | 87
participants | 31 | 31
Statistical Analysis 1: Comparison: Bangerter vs Patching; Logistic regression was used to compare the proportion of patients with 3 or more lines of amblyopic eye visual acuity improvement from baseline to 24 weeks; Test type: Superiority or Other; p = 0.61, Regression, Logistic

9. Secondary Outcome: Distribution of Patient Characteristics at the 24-week Outcome Exam.
Description: The distribution of the number of participants in each patient characteristic category at the 24-week outcome examination was found (for example, the number of participants at 24 weeks who were 3 to <5 years old at the time of enrollment).
Time Frame: 24 weeks
Measure: Number; unit: participants
Arm/Group | Bangerter | Patching
Number analyzed (Participants) | 81 | 88
participants
  Female | 34 | 43
  Male | 47 | 45
  White, non-Hispanic | 63 | 61
  Non-white or Hispanic | 17 | 26
  Age at enrollment: 3 to <5 yrs | 21 | 23
  Age at enrollment: 5 to <7 yrs | 31 | 34
  Age at enrollment: 7 to <10 yrs | 29 | 31
  Prior treatment for amblyopia: No | 65 | 75
  Prior treatment for amblyopia: Yes | 16 | 13
  Cause of amblyopia: Strabismus | 21 | 23
  Cause of amblyopia: Anisometropia | 36 | 39
  Cause of amblyopia: Strabismus and anisometropia | 24 | 26
  Distance VA in amblyopic eye: 20/80 (worse) | 15 | 22
  Distance VA in amblyopic eye: 20/63 | 25 | 29
  Distance VA in amblyopic eye: 20/50 | 20 | 17
  Distance VA in amblyopic eye: 20/40 (best) | 21 | 20

10. Secondary Outcome: Mean and SD of Change in Visual Acuity in the Amblyopic Eye From Baseline to 24-Week Outcome Examination According to Patient Characteristics
Description: as for outcome 4
Time Frame: Baseline to 24 weeks
Measure: Mean (Standard Deviation); unit: logMAR line
Arm/Group | Bangerter | Patching
Number analyzed (Participants) | 81 | 88
logMAR line
  Female | 2.1 (1.7) | 2.4 (1.3)
  Male | 1.7 (1.6) | 2.2 (1.3)
  White, non-Hispanic | 1.8 (1.7) | 2.3 (1.3)
  Non-white or Hispanic | 2.1 (1.4) | 2.4 (1.3)
  Age at enrollment: 3 to <5 yrs | 2.1 (1.9) | 2.7 (1.4)
  Age at enrollment: 5 to <7 yrs | 2.1 (1.7) | 2.5 (1.2)
  Age at enrollment: 7 to <10 yrs | 1.5 (1.3) | 1.8 (1.2)
  Prior treatment for amblyopia: No | 1.9 (1.7) | 2.4 (1.3)
  Prior treatment for amblyopia: Yes | 2.0 (1.4) | 1.7 (1.0)
  Cause of amblyopia: Strabismus | 2.2 (1.5) | 2.4 (1.3)
  Cause of amblyopia: Anisometropia | 1.5 (1.7) | 2.4 (1.4)
  Cause of amblyopia: Strabismus and anisometropia | 2.2 (1.5) | 2.1 (1.2)
  Distance VA in amblyopic eye: 20/80 (worse) | 2.3 (2.0) | 2.3 (1.3)
  Distance VA in amblyopic eye: 20/63 | 1.8 (1.7) | 2.5 (1.5)
  Distance VA in amblyopic eye: 20/50 | 1.7 (1.7) | 2.3 (1.4)
  Distance VA in amblyopic eye: 20/40 (best) | 1.9 (1.0) | 2.0 (1.1)

11. Secondary Outcome: Distribution of Change in Randot Preschool Stereoacuity From Baseline to 24-Week Outcome by Treatment Group: All Subjects
Description: The Randot Preschool Stereotest measures stereopsis from 800 to 40 seconds of arc. It is designed as a matching game in which the patient matches pictures in a test booklet wearing special glasses. A subject can fail the pretest (not see any pictures) or can score >800 (the worst), 800, 400, 200, 100, 60, or 40 (the best). If two shapes are identified correctly the patient moves to the next lower level. A failed test occurs when the patient cannot identify any shapes. A change of 1 level is a movement of 1 step in the scale (decrease shows improvement - ex. 100 to 60 is 1 level improved).
Time Frame: Baseline to 24 weeks
Measure: Number; unit: participants
Arm/Group | Bangerter | Patching
Number analyzed (Participants) | 76 | 80
participants
  >=2 levels improved | 12 | 15
  Within 1 level | 61 | 58
  >=2 levels worsened | 3 | 7
Statistical Analysis 1: Comparison: Bangerter vs Patching; A Wilcoxon rank-sum test was used to evaluate change in Randot Preschool stereoacuity levels from baseline to 24 weeks by treatment group; Test type: Superiority or Other; p = 0.90, Wilcoxon rank-sum

12. Secondary Outcome: Distribution of Change in Randot Preschool Stereoacuity From Baseline to 24-week Outcome by Treatment Group: Subjects With Anisometropia and No Strabismus
Description: as for outcome 11
Time Frame: Baseline to 24 weeks
Measure: Number; unit: participants
Arm/Group | Bangerter | Patching
Number analyzed (Participants) | 33 | 34
participants
  >=2 levels improved | 7 | 9
  Within 1 level | 25 | 21
  >=2 levels worsened | 1 | 4
Statistical Analysis 1: Comparison: Bangerter vs Patching; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.88, Wilcoxon rank-sum

13. Secondary Outcome: Distribution of Change in Fellow Eye Visual Acuity From Baseline to 24 Weeks
Description: as for outcome 4
Time Frame: Baseline to 24 weeks
Measure: Number; unit: participants
Arm/Group | Bangerter | Patching
Number analyzed (Participants) | 81 | 88
participants
  3 lines or worse | 0 | 0
  2 lines worse | 1 | 5
  1 line worse | 17 | 8
  0 lines | 39 | 40
  1 line better | 20 | 23
  2 lines better | 4 | 11
  3 lines or better | 0 | 1

14. Secondary Outcome: Mean Change in Fellow Eye Visual Acuity From Baseline to 24 Weeks
Description: as for outcome 4
Time Frame: Baseline to 24 weeks
Measure: Mean (Standard Deviation); unit: logMAR line
Arm/Group | Bangerter | Patching
Number analyzed (Participants) | 81 | 88
logMAR line | 0.09 (0.84) | 0.36 (1.1)
Statistical Analysis 1: Comparison: Bangerter vs Patching; A treatment group difference in the fellow eye visual acuity at 24 weeks was evaluated in an ANCOVA model adjusted for the baseline fellow eye acuity; Test type: Superiority or Other; p = 0.07, ANCOVA
Statistical Analysis 2: Comparison: Bangerter vs Patching; The Fisher exact test was used to compare the proportion of subjects in each treatment group who tested 2 or more logMAR lines worse in the fellow eye at 24 weeks compared with baseline; Test type: Superiority or Other; p = 0.21, Fisher Exact

15. Secondary Outcome: Impact of Treatment on Patient and Family at 6 Weeks
Description: The Parental Amblyopia Treatment Index consists of 18 likert-type questions evaluating the impact of treatment on the patient and family. Questions are answered on a scale from 'Strongly Disagree' to 'Strongly Agree.' For analysis, values were coded numerically with integers from 5 (strongly agree) to 1 (strongly disagree) (0 was assigned to 'non-applicable' answers). The scores were summed and averaged for each individual (total sums could range from 0 to 90; means could range from 0 to 5). A mean across all individuals was computed from the individual means.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Bangerter | Patching
Number analyzed (Participants) | 79 | 81
Units on a scale | 2.1 (1.1) | 2.3 (1.0)
Statistical Analysis 1: Comparison: Bangerter vs Patching; A t-test was used to evaluate treatment group difference of impact of treatment at 6 weeks; Test type: Superiority or Other; p = 0.03, t-test, 2 sided

16. Secondary Outcome: Impact of Treatment on Patient and Family at 24 Weeks
Description: as for outcome 15
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Bangerter | Patching
Number analyzed (Participants) | 75 | 75
Units on a scale | 1.9 (1.0) | 2.3 (1.1)
Statistical Analysis 1: Comparison: Bangerter vs Patching; A t-test was used to evaluate treatment group difference of impact of treatment at 24 weeks; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

17. Secondary Outcome: Adverse Effects of Treatment on Patient and Family at 6 Weeks
Description: The Parental Amblyopia Treatment Index consists of 18 likert-type questions evaluating the impact of treatment on the patient and family (8 of these questions pertain to adverse effects of treatment). Questions are answered on a scale from 'Strongly Disagree' to 'Strongly Agree.' For analysis, values were coded numerically with integers from 5 (strongly agree) to 1 (strongly disagree) (0 was assigned to 'non-applicable' answers). The scores for these 8 questions were summed and averaged for each individual (total sums could range from 0 to 40). A mean across all individuals was computed.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Bangerter | Patching
Number analyzed (Participants) | 79 | 81
Units on a scale | 2.2 (0.7) | 2.2 (0.6)
Statistical Analysis 1: Comparison: Bangerter vs Patching; A t-test was used to evaluate treatment group difference of the adverse effects subscale at 6 weeks; Test type: Superiority or Other; p = 0.90, t-test, 2 sided

18. Secondary Outcome: Adverse Effects of Treatment on Patient and Family at 24 Weeks
Description: as for outcome 17
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Bangerter | Patching
Number analyzed (Participants) | 75 | 75
Units on a scale | 1.9 (0.7) | 2.2 (0.6)
Statistical Analysis 1: Comparison: Bangerter vs Patching; A t-test was used to evaluate treatment group difference of the adverse effects subscale at 24 weeks; Test type: Superiority or Other; p = 0.01, t-test, 2 sided

19. Secondary Outcome: Compliance With Treatment at 6 Weeks
Description: The Parental Amblyopia Treatment Index consists of 18 likert-type questions evaluating the impact of treatment on the patient and family (7 of these questions pertain to compliance of treatment). Questions are answered on a scale from 'Strongly Disagree' to 'Strongly Agree.' For analysis, values were coded numerically with integers from 5 (strongly agree) to 1 (strongly disagree) (0 was assigned to 'non-applicable' answers). The scores for these 7 questions were summed and averaged for each individual (total sums could range from 0 to 35). A mean across all individuals was computed.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Bangerter | Patching
Number analyzed (Participants) | 79 | 81
Units on a scale | 2.3 (1.0) | 2.5 (0.8)
Statistical Analysis 1: Comparison: Bangerter vs Patching; A t-test was used to evaluate treatment group difference of the compliance subscale at 6 weeks; Test type: Superiority or Other; p = 0.12, t-test, 2 sided

20. Secondary Outcome: Compliance With Treatment at 24 Weeks
Description: as for outcome 19
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Bangerter | Patching
Number analyzed (Participants) | 75 | 75
Units on a scale | 2.1 (0.9) | 2.6 (0.9)
Statistical Analysis 1: Comparison: Bangerter vs Patching; A t-test was used to evaluate treatment group difference of the compliance subscale at 24 weeks; Test type: Superiority or Other; p = 0.001, t-test, 2 sided

21. Secondary Outcome: Social Stigma From Treatment at 6 Weeks
Description: The Parental Amblyopia Treatment Index consists of 18 likert-type questions evaluating the impact of treatment on the patient and family (2 of these questions pertain to social stigma of treatment). Questions are answered on a scale from 'Strongly Disagree' to 'Strongly Agree.' For analysis, values were coded numerically with integers from 5 (strongly agree) to 1 (strongly disagree) (0 was assigned to 'non-applicable' answers). The scores for these 2 questions were summed and averaged for each individual (total sums could range from 0 to 10). A mean across all individuals was computed.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Bangerter | Patching
Number analyzed (Participants) | 79 | 81
Units on a scale | 1.7 (0.6) | 2.4 (0.9)
Statistical Analysis 1: Comparison: Bangerter vs Patching; A t-test was used to evaluate treatment group difference of social stigma at 6 weeks; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

22. Secondary Outcome: Social Stigma From Treatment at 24 Weeks
Description: as for outcome 21
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Bangerter | Patching
Number analyzed (Participants) | 75 | 75
Units on a scale | 1.6 (0.7) | 2.4 (0.8)
Statistical Analysis 1: Comparison: Bangerter vs Patching; A t-test was used to evaluate treatment group difference of social stigma at 24 weeks; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Patching | Bangerter Filters
Serious Adverse Events (participants affected / at risk) | 0/97 | 0/89
Other Adverse Events (participants affected / at risk) | 0/97 | 0/89

LIMITATIONS AND CAVEATS:
Compliance assessment was based on parents' diaries and judgment by the researchers. Because we did not use an objective method to measure occlusion or spectacle wear, we cannot guarantee that the patients adhered to their prescribed regimens.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No